CLINICAL TRIAL: NCT07328165
Title: Core Stability vs Respiratory Muscle Training in Children With Down Syndrome
Brief Title: The Impact of Core Stability Versus Respiratory Muscle Strengthening Exercises on Bone Mineral Density in Children With Down Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Saeed Alsakhawi, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005953
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Down Syndrome (DS); Low Bone Mineral Density
MeSH Terms: conditions — Down Syndrome; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core Stability Exercise Group (Experimental): This group will receive core stability exercises in addition to physical therapy program as control group.
  Interventions: Behavioral: Core Stability Exercise Group
- Respiratory Muscle Strengthening Group (Experimental): This group will receive respiratory muscle strengthening exercises in addition to physical therapy program as control group
  Interventions: Device: Respiratory Muscle Strengthening Group
- Control Group (Active Comparator): The control group will receive the physical therapy program and conduct three times peer week over 8 consecutive weeks under the supervision of a physical rehabilitation specialist
  Interventions: Behavioral: Control /Conventional Physiotherapy Group

INTERVENTIONS:
Behavioral: Core Stability Exercise Group — Based on Jeffrey's protocol, the protocol includes specific spinal stabilization exercises, lumbar-pelvic proprioception retraining, and abdominal maneuvers (holding the abdomen in) and multifidus muscle contraction, followed by maintaining stabilization maneuver using dynamic stability achieved in different positions (supine, prone, and squatting) and addition of dynamic elements (limb movement, use of Swiss ball) in later stages.
  Arms: Core Stability Exercise Group
Device: Respiratory Muscle Strengthening Group — By using a threshold inspiratory muscle training (IMT) (Respironics, Cedar Grove, NJ, USA). Frequency 3 time per week for 8 weeks. It is a spring-loaded valve that inspiratory resistance can be adjusted. This training last for 30 min. To develop muscle strength; during the first 10 min of practice, threshold IMT will be used in 10 series of 60s each, separated by rest periods of 60s. To develop endurance; during the final 20 min, the equipment will be used uninterruptedly. Prior to the beginning of each session, the pressure threshold load throughout the practice will be 50 % of Maximum Inspiratory pressure that will be calculated during the evaluation of children.
  Arms: Respiratory Muscle Strengthening Group
Behavioral: Control /Conventional Physiotherapy Group — The primary focus of the program was to improve bone mineral density. Each session will be conducted 60 minutes and consist of weight bearing exercises and strengthen exercises in the form of isometric exercises;
  Arms: Control Group

SUMMARY:
Children with Down syndrome often exhibit diminished physical fitness levels and lower bone mass. Numerous factors contribute to this decrease in bone mass density, including decreased levels of leptin, reduced muscle mass and strength, impaired balance, and skeletal abnormalities. These factors further exacerbate the risk of developing osteoporosis in this population. Therefore, it is crucial to prioritize interventions that focus on maximizing peak bone mass during childhood in order to enhance the quality of life for adults with Down syndrome. The study aims to compare the impact of core stability exercises and respiratory muscle strengthening exercises on bone mineral density in children with Down syndrome. Sixty Children with Down syndrome will be assessed and included in this study. The age of children will range from 10 to 13 years. Children will be allocated randomly into three groups (control and two study group A & B). The control group receives a physical therapy program, study group A receives traditional physical therapy program with core stability exercises, and study group B receives traditional physical therapy program with respiratory muscle strengthening exercises. Groups will be evaluated using dual energy X-ray absorptiometry DXA (DPX-IQ, version 4.6A). Bone mineral density (BMD) of femoral neck and lumbar spine will be determined and the mean density will be expressed as g/cm2.

ELIGIBILITY:
Inclusion Criteria:

* Age will range from 10-13 years
* Diagnosed with Down syndrome.
* Children with the ability to understand and follow verbal commands and instructions used during training and tests
* Able to stand and walk independently

Exclusion Criteria:

* Any neurological, mobility disorders, vision or hearing loss, cardiac anomalies or musculoskeletal disorder
* With asthma or any chronic chest diseases
* With significant tightness or deformities in the lower limbs and limber spine

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density (BMD) of femoral neck and lumbar spine | 8 weeks
  . Groups will be evaluated using dual energy X-ray absorptiometry DXA (DPX-IQ, version 4.6A).